CLINICAL TRIAL: NCT01268111
Title: Effect of Vitamin D Supplementation on Insulin Sensitivity and Retinol-binding Protein 4 Levels in Subjects With Vitamin D Deficiency
Brief Title: Effect of Vitamin D Replacement on Insulin Sensitivity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TTUHSC-VitD-RBP4
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Insulin Sensitivity
Keywords: vitamin D deficiency, insulin sensitivity
MeSH Terms: conditions — Insulin Resistance; Vitamin D Deficiency | interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): ERgocalcifoerol 50,000 units q weekly for 8 weeks
  Interventions: Drug: Ergocalciferols
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergocalciferols — ERgocaclciferol 50,000 units weekly for 8 weeks
  Arms: Vitamin D
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
Healthy subjects with low Vitamin D levels will be randomly assigned to either Vitamin D replacement or placebo for a period of 8 weeks. Insulin sensitivity will be measured before and after the intervention, and the changes will be compared between the two groups. This will help us understand if Vitamin D replacement improves insulin sensitivity. Serum Retinol Binding Protein 4 levels will also be measured to see if changes in insulin sensitivity are mediated by RBP4.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-60 years 2. No known medical illnesses requiring pharmacotherapy 3. Not on any mineral or vitamin supplements in the last 3 months

Exclusion Criteria:

* 1. Subjects requiring prompt initiation of pharmacotherapy, such as those with incidentally discovered diabetes mellitus or hypertension.

  2. Previous administration of glucocorticoids, retinoic acid derivatives, or insulin sensitizers in the preceding 3 months.

  3. Bariatric surgery or liposuction 4. Unintentional weight loss >5% of the body weight in last 3 months 5. Chronic smokers (> 1 pk/d for 10 years) 6. Alcohol use > 2 drinks/day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinaya Simha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Texas Tech University Health Sciences Center, Odessa, Texas, United States

REFERENCES:
- [Result] Simha V, Mahmood M, Ansari M, Spellman CW, Shah P. Effect of vitamin D replacement on insulin sensitivity in subjects with vitamin D deficiency. J Investig Med. 2012 Dec;60(8):1214-8. doi: 10.2310/JIM.0b013e3182747c06. PMID 23111651

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo q weekly for 8 weeks
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (3.6) | 27.8 (2.6) | 28.4 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: M Value (Insulin Stimulated Glucose Uptake)
Description: Insulin stimulated glucose uptake will be measured by glucose clamp studies
Time Frame: Baseline and at 8 weeks
Measure: Mean (Standard Deviation); unit: mg/kg.min
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 6 | 6
mg/kg.min
  Baseline | 4.1 (1.56) | 5.6 (1.48)
  8 weeks | 4.7 (1.35) | 5.5 (1.68)
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority or Other; p = 0.4, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Vitamin D | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes